CLINICAL TRIAL: NCT06912269
Title: Effects of Strength Training at Different Intensities on the Plantar Flexors' Functional, Neuromuscular, and Tendon Properties After Achilles Tendon Rupture
Brief Title: Effects of Strength Training on the Plantar Flexors' Properties After Achilles Tendon Rupture
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Jeam Marcel Geremia, Principal Investigator, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6786944
Record Dates: First submitted 2024-10-10; First posted 2025-04-04 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Achilles Tendon Rupture; Strength Training Adaptations; Neuromuscular Adaptations
Keywords: Neuromuscular plasticity; Stiffness; Functionality; Triceps surae; Calcaneal tendon rupture
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Strength training (low intensity) (Experimental): Twelve weeks of strength training program for the calf muscles, with low load intensity
  Interventions: Other: Exercise
- Strength training (moderate intensity) (Experimental): Twelve weeks of strength training program for the calf muscles, with moderate load intensity
  Interventions: Other: Exercise
- Healthy subjects (No Intervention): A control condition composed of healthy individuals (i.e., without any injury), who will not receive any training, will be used as a comparison at the beginning and end of the intervention.

INTERVENTIONS:
Other: Exercise — A progressive calf strength training program lasting 12 weeks (twice weekly sessions), with a total of 25 visits to the gym. Specific exercises for ankle flexors: standing unilateral plantar flexion (on the machine) and seated unilateral plantar flexion (adapted on the Smith machine) will be performed. Participants will use progressive load from 55% of one repetition maximum load for the specific plantar flexion exercises.
  Arms: Strength training (low intensity)
Other: Exercise — A progressive calf strength training program lasting 12 weeks (twice weekly sessions), with a total of 25 visits to the gym. Specific exercises for ankle flexors: standing unilateral plantar flexion (on the machine) and seated unilateral plantar flexion (adapted on the Smith machine) will be performed. Participants will use progressive load from 70% of one repetition maximum load for the specific plantar flexion exercises.
  Arms: Strength training (moderate intensity)

SUMMARY:
Among the injuries that affect the Achilles tendon, rupture is one of the most frequent. This injury can generate functional, neuromuscular, and tendon deficits that can last for long periods or even be permanent. In the long term (i.e., more than a year after the injury), individuals present functional impairments related to the lower limb, deficits in the capacity to produce muscle force, as well as higher levels of muscle activation (as a compensatory response). Such changes may be due to injury adaptations in the plantar flexor muscles' architecture, which may have shorter, more pennate fibers, leading to reduced muscle thickness. Furthermore, the Achilles tendon may be elongated, with a greater cross-sectional area, presenting lower stiffness and quality (i.e., lower Young's modulus). Strength training can play an important role in recovering from Achilles tendon ruptures, as it promotes functional, neuromuscular, and tendon adaptations that can minimize deficits caused by the injury. However, there is a gap in the literature regarding strength training, as well as the dose vs response relationship, regarding functional, neuromuscular, and tendon adaptations after Achilles tendon rupture. Thus, the aim of the present study is to compare the effects of a strength training program of different intensities on plantar flexors' functional, neuromuscular, and tendon outcomes after Achilles tendon rupture. Men aged between 20 and 50 years old who suffered a total unilateral rupture of the Achilles tendon between one and five years after the rupture will be included in the study, as well as healthy men who did not suffer the rupture (control group). Participants who have suffered an Achilles tendon rupture will undergo a progressive lower limb strength training program twice a week for a total duration of 12 weeks, which will be randomized between two groups: low intensity (G55 - 55% of 1-RM) and moderate intensity (G70 - 70% of 1-RM). The following outcomes will be evaluated: a) Achilles tendon's morphological (length and cross-sectional area), mechanical (force-elongation relationship and stiffness) and material (stress-strain relationship and Young's modulus) properties; b) triceps surae muscles' morphological (architecture [fascicle length, pennation angle and thickness] and quality [measured by echointensity and specific tension]) properties; c) ankle functionality (maximum height in the heel raise test); d) the plantar flexors' force production capacity (peak and rate of torque development in different joint positions); e) the plantar flexors' muscle voluntary activation; and f) triceps suraes' neuromuscular capacity (i.e., recruitment curves). Assessments will be performed at two times (pre-training; and after 12 weeks of training [post-12]) through functional tests, ultrasound techniques, isokinetic dynamometry, electromyography, and percutaneous electrical stimulation. An intraclass correlation coefficient will be used to verify the test-retest reproducibility of ultrasound measurements. The Chi-Square test will be used to compare the level of physical activity (pre-training) between the groups. The results of the intervention will be expressed using descriptive statistics (mean, standard deviation, and standard error). The normality and sphericity of the data will be tested using the Shapiro-Wilk and Mauchly tests, respectively. A generalized estimating equation, followed by Bonferroni post-hoc, will be used to compare the effects of groups (G55 and G70) and times (pre-training, Post-6, and Post-12). A one-way ANOVA, followed by a Bonferroni post-hoc, will be used to compare the control group participants' limbs with the healthy and injured limbs from both intervention groups (G55 and G70) in the Pre and Post-12 times. The effect size will be estimated for each outcome. All statistical analyzes will be performed using SPSS software.

DETAILED DESCRIPTION:
Among the injuries that affect the Achilles tendon, rupture is one of the most frequent. This injury can generate functional, neuromuscular, and tendon deficits that can last for long periods or even be permanent. In the long term (i.e., more than a year after the injury), individuals present functional impairments related to the lower limb, deficits in the capacity to produce muscle force, as well as higher levels of muscle activation (as a compensatory response). Such changes may be due to injury adaptations in the plantar flexor muscles' architecture, which may have shorter, more pennate fibers, leading to reduced muscle thickness. Furthermore, the Achilles tendon may be elongated, with a greater cross-sectional area, presenting lower stiffness and quality (i.e., lower Young's modulus). Strength training can play an important role in recovering from Achilles tendon ruptures, as it promotes functional, neuromuscular, and tendon adaptations that can minimize deficits caused by the injury. However, there is a gap in the literature regarding strength training, as well as the dose vs response relationship, regarding functional, neuromuscular, and tendon adaptations after Achilles tendon rupture. Thus, the aim of the present study is to compare the effects of a strength training program of different intensities on plantar flexors' functional, neuromuscular, and tendon outcomes after Achilles tendon rupture. Men aged between 20 and 50 years old who suffered a total unilateral rupture of the Achilles tendon between one and five years after the rupture will be included in the study, as well as healthy men who did not suffer the rupture (control group). Participants who have suffered an Achilles tendon rupture will undergo a progressive lower limb strength training program twice a week for a total duration of 12 weeks, which will be randomized between two groups: low intensity (G55 - 55% of 1-RM) and moderate intensity (G70 - 70% of 1-RM). The following outcomes will be evaluated: a) Achilles tendon's morphological (length and cross-sectional area), mechanical (force-elongation relationship and stiffness) and material (stress-strain relationship and Young's modulus) properties; b) triceps surae muscles' morphological (architecture [fascicle length, pennation angle and thickness] and quality [measured by echointensity and specific tension]) properties; c) ankle functionality (maximum height in the heel raise test); d) the plantar flexors' force production capacity (peak and rate of torque development in different joint positions); e) the plantar flexors' muscle voluntary activation; and f) triceps suraes' neuromuscular capacity (i.e., recruitment curves). Assessments will be performed at two times (pre-training; and after 12 weeks of training [post-12]) through functional tests, ultrasound techniques, isokinetic dynamometry, electromyography, and percutaneous electrical stimulation. An intraclass correlation coefficient will be used to verify the test-retest reproducibility of ultrasound measurements. The Chi-Square test will be used to compare the level of physical activity (pre-training) between the groups. The results of the intervention will be expressed using descriptive statistics (mean, standard deviation, and standard error). The normality and sphericity of the data will be tested using the Shapiro-Wilk and Mauchly tests, respectively. A generalized estimating equation, followed by Bonferroni post-hoc, will be used to compare the effects of groups (G55 and G70) and times (pre-training, Post-6, and Post-12). A one-way ANOVA, followed by a Bonferroni post-hoc, will be used to compare the control group participants' limbs with the healthy and injured limbs from both intervention groups (G55 and G70) in the Pre and Post-12 times. The effect size will be estimated for each outcome. All statistical analyzes will be performed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 18 to 64 who have ruptured their Achilles tendon unilaterally no more than 5 years ago;
* Who are not performing systematic and regular calf strength training.

Exclusion Criteria:

* Non-surgical treatment for Achilles tendon rupture;
* History of postsurgical complications (infection or re-rupture);
* Presence of any type of ankle injury in the last six month;
* Participation in a strength training program for plantar flexors in the last six months prior to participation in the study;
* Having heart failure; autoimmune diseases; and/or diabetes;
* Systematic use of antibiotics or steroids within the last 12 months;
* Presence of any other clinical contraindication for performing maximum strength tests.

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Changes in foot and ankle joint function | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  The foot and ankle joint function will be assessed through Foot and Ankle Outcome Score, which evaluate five different domains: pain, other symptoms, activities of daily living, sports and recreational activities, and quality of life related to the ankle and foot.
Changes in Achilles tendon function and symptom | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Achilles tendon post-rupture function and symptoms will be assessed through Achilles Tendon Rupture Score (ATRS).
Changes in ankle functional performance | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  The ankle functional performance will be assessed using the heel raise test. With this test, the maximum height of the heel lift will be assessed, corresponding to the measurement of functionality of the ankle plantar flexors.
Changes in plantar flexors' muscle strength | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  The plantar flexors' muscle strength will be assessed by the peak torque in different ankle joints (i.e., -10º, 0º, and 20º of plantar flexion - 0º neutral position).
Changes in Achilles tendon stiffness | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Tendon stiffness will be obtained by calculating the slope in the last 10% of the linear region of the force-deformation curve.

SECONDARY OUTCOMES:
Changes in Achilles tendon Young's Modulus | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Tendon stiffness will be obtained by calculating the slope in the last 10% of the linear region of the stress-strain curve.
Changes in Achilles tendon morphological properties | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Tendon morphological properties will be obtained by the total tendon length (distance between medial gastrocnemius muscle-tendon junction and tendon distal insertion in the calcaneous bone), free tendon length (soleus muscle-tendon junction and tendon distal insertion), and tendon's cross sectional area (measured at 2, 4, and 6cm from the tendon distal insertion).
Changes in plantar flexors' muscle arquitecture | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  The muscular architecture of the plantar flexor muscles will be evaluated using B-mode ultrasound images. Imagem analyses will be performed to identify the pennation angle and length of the muscle fascicles, and the muscle thickness of each triceps surae muscle.
Changes in plantar flexors' muscle activation | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Muscle activation will be captured during muscle voluntary isometric contraction (MVIC) testes, at different joint positions. The maximum root mean square (RMS) values of each plantar flexor muscle will be calculated for each of the MVICs produced during the isometric peak torque assessments. These RMS values will be obtained by means of 1-s duration cuts (corresponding to 2000 points) of the MVICs during the torque signal plateau.
Changes in neuromuscular recruitment capacity | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  Muscle activation parameters evoked by percutaneous neuromuscular electrical stimulation techniques will be obtained through neuromechanical responses. Recruitment curves will be constructed to evaluate the neuromuscular capacity of the plantar flexors, based on the peak-to-peak amplitudes of the M waves and H reflexes, which will be mapped and recorded simultaneously.

OTHER OUTCOMES:
Changes in plantar flexors' muscle power | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  The torque values obtained during the maximal voluntary isometric contractions (MVICs) tests will be used to determine the peak torque, as well as for the analysis of the rate of torque development (RTD). The active torque values produced in the torque-time curve obtained during the MVICs will allow the analysis of the RTD, which will be calculated in each joint position from the derivative of the torque-time curve (Nm s-1), from the beginning of the contraction (onset = 0-ms) to 50, 100, 200 and 400-ms, in addition to the interval between 200 and 400-ms.
Changes in plantar flexors' muscle quality | From baseline measurements up to 13 weeks after (i.e., one week after the end of the training program)
  In addition to the analysis of the muscle architecture, the images obtained for each plantar flexor muscle will allow the simultaneous analysis of the muscle quality measured by echointensity. During this analysis, the region of interest that includes the largest muscle area between the deep and superficial aponeuroses (avoiding wrapping tissues and bone) will be considered, for which the mean values of a histogram corresponding to the values in gray scale [scale from 0 (black) to 255 (white)] will be calculated. In addition, muscle quality will also be estimated by specific tension, expressed as force/torque per unit of muscle mass, which will be calculated by the ratio between the peak torque of the plantar flexors, obtained during isometric tests with the ankle in the neutral position (i.e., 0º of plantar flexion), and the amount of muscle mass representative of the triceps surae.

CONTACTS AND LOCATIONS:
Overall Officials: Jeam M Geremia, PhD, Study Director — Federal University of Rio Grande do Sul; Marcelo H Glänzel, MSc, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Exercise Research Laboratory (LAPEX) - School of Physical Education, Physiotherapy, and Dance, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided